CLINICAL TRIAL: NCT06819033
Title: Effects of Photobiomodulation on Pain After Presentation of Aphthous Ulcers in Pediatric Dental Patients
Brief Title: Effects of Photobiomodulation (PBM) on Pain After Presentation of Aphthous Ulcers in Pediatric Dental Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Brett Thomas Chiquet, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-DB-24-1153
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Aphthous Ulcer
Keywords: magic mouthwash; laser treatment
MeSH Terms: conditions — Stomatitis, Aphthous | interventions — Low-Level Light Therapy; aluminum hydroxide, magnesium hydroxide, drug combination; Diphenhydramine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- PBM Therapy (Experimental)
  Interventions: Device: PBM Therapy; Drug: Maalox plus Benadryl
- Standard of care (Active Comparator)
  Interventions: Drug: Maalox plus Benadryl

INTERVENTIONS:
Device: PBM Therapy — patients will receive PBM therapy using the Biolase Epic pro laser. An average power of 0.6w (peak power = 80w, rep. rate= 20Hz). Each aphthous ulcer will be irradiated one time for a total of 30 seconds via continuous wave.
  Arms: PBM Therapy
Drug: Maalox plus Benadryl — 1:1 mixture of Maalox and Benadryl will be applied to the ulcer as needed for pain. Applications typically will be applied before eating to form a dissolvable oral band-aid that lasts for up to 30 minutes. 10 milliliters of 1:1 Maalox: Benadryl solution will be provided to the family. During the presenting appointment, the patient/family will be shown how to use the 1:1 Maalox: Benadryl solution. It will be applied topically with no rinsing needed.

SUMMARY:
The purpose of this study is to compare the efficacy of laser photobiomodulation and "Magic Mouthwash" for treatment of pain in pediatric patients with aphthous ulcers , to assess how photobiomodulation influences the rate of healing of aphthous ulcers in pediatric patients and to measure changes in pain levels reported by pediatric patients undergoing photobiomodulation treatment for aphthous ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Patient/guardian speaks either English or Spanish
* Patient presenting with one or more aphthous ulcers in their mouth, identified during a scheduled dental appointment
* No previous PBM treatment to the presenting aphthous ulcer(s)
* Guardian able to partake in a follow-up phone call in either the English or Spanish language

Exclusion Criteria:

* Patient presents with aphthous ulcers recently treated with PBM
* Patient presents with herpes labialis (cold sores)
* Patients presents with systemic disease that affects soft tissue/mucous healing

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of life as assessed by questionnaire (Likert scale) | Baseline, immediately after treatment(about 5 minutes), 24 hours after treatment
  This is a 6 item questionnaire and each is scored from 1-5, maximum score of 30,higher number indicating better outcome
Pain as assessed by how frequently patient complains of pain (Likert scale) | upto 24 hours after treatment
Pain as assessed by number of participants who are using any over-the-counter or prescription medications, topical treatments, or oral rinses to treat aphthous ulcer pain | upto 24 hours after treatment

SECONDARY OUTCOMES:
Change in lesion size as an indication of healing as assessed by clinical intraoral images of the aphthous ulcer and measuring tool | pre-treatment and immediately post-treatment(about 5 minutes)
Change in pain as assessed by a Visual Analogue Scale (VAS) for control group | Baseline, 24 hours after treatment
  Pain level is scored from 0(no pain) to 10(worst pain)
Pain as assessed by a Visual Analogue Scale (VAS) for experimental group | Baseline, immediately after PBM(about 5 minutes), 24 hours after treatment
  Pain level is scored from 0(no pain) to 10(worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Chiquet, DDS, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No